CLINICAL TRIAL: NCT04136977
Title: XprESS Eustachian Tube Balloon Dilation Registry
Brief Title: XprESS ET Registry
Status: Completed | Type: Observational
Sponsor: Entellus Medical, Inc. (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Other Study IDs: 4079-001
Record Dates: First submitted 2019-10-02; First posted 2019-10-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Eustachian tube dilation — Unilateral or bilateral balloon dilation of the Eustachian tube using the FDA-cleared XprESS ENT Dilation System
  Other Names: XprESS ET balloon dilation

SUMMARY:
A prospective, multicenter, registry of patients undergoing balloon dilation of the Eustachian tubes (ET).

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, postmarket registry enrolling up to 300 participants who are planning to undergo balloon dilation of the Eustachian tubes for treatment of chronic/persistent Eustachian tube dysfunction (ETD). Procedural information will be collect as well as efficacy and safety data through 6 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have been diagnosed with persistent/chronic Eustachian tube dysfunction (duration 3 months or more)
* Be a candidate for unilateral or bilateral Eustachian tube balloon dilation using the XprESS device
* Be able to read and understand English
* Be willing and able to provide informed consent
* Be willing to comply with the protocol requirements

Exclusion Criteria:

* Have a history of patulous Eustachian tube
* Require additional ear surgery (eg, myringotomy, tympanostomy) at the time of study procedure
* Have evidence of internal carotid artery dehiscence
* Be currently participating in any other drug or device clinical studies, excluding postapproval or marketing registry studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with persistent/chronic Eustachian tube dysfunction who are undergoing balloon dilation of the Eustachian tubes.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Change in mean Eustachian Tube Dysfunction Questionnaire (ETDQ-7) score | 6 Months
  Change from baseline to follow-up in the mean overall ETDQ-7 score. The ETDQ-7 is a validated 7-item patient-reported questionnaire reporting the presence and severity of symptoms associated with Eustachian tube dysfunction. Each item is scored from 1 (normal) to 7 (severe). The overall score is the mean score of the 7 items.
Complication rate | 6 Months
  Percentage of participants who experience 1 or more serious adverse events that are related to the device and/or procedure.

SECONDARY OUTCOMES:
Procedural information | Procedure through 6-week follow-up
  Details of the balloon dilation procedure, including setting, anesthesia, technical success, concomitant procedures, procedure/device-related adverse events, and recovery time.
Minimal clinically important difference in ETDQ-7 score | 6 Months
  Percentage of participants achieving the minimal clinical important difference in overall ETDQ-7 score (reduction from baseline of 0.5 points or more). The ETDQ-7 is a validated 7-item patient-reported questionnaire reporting the presence and severity of symptoms associated with Eustachian tube dysfunction. Each item is scored from 1 (normal) to 7 (severe). The overall score is the mean score of the 7 items.
Revision Eustachian tube dilation | 6 Months
  Percentage of participants who require revision dilation on an ear that was treated in the initial procedure.
Surgical interventions | 6 Months
  Percentage of participants requiring surgical ear intervention (other than balloon dilation) on an ear that was treated in the initial procedure but has recurrent or continuing ETD symptoms.
Participant satisfaction: Proportion of participants indicating satisfaction and willing to recommend the procedure to friends or family | 6 Months
  Percentage of participants indicating satisfaction and willing to recommend the procedure to friends or family.
Change in work productivity/activity impairment | 6 Months
  Participants complete the validated Work Productivity and Activity Impairment (WPAI) at baseline and 6 month follow-up. The questionnaire consists of 6 questions that evaluate absenteeism, presenteeism, work productivity loss, and activity impairment over the previous week. Results are expressed as the percentage of impairment from 0 to 100, for which higher numbers indicate worse outcomes (ie, greater impairment and less productivity). Absenteeism is calculated by dividing the number of hours missed by the sum of the numbers of hours missed plus the number of hours worked. Presenteeism, is calculated by dividing the response to productivity at work question by 10, while activity impairment is calculated by dividing the response to the ability to carry out daily activities question by 10. Finally, the overall work impairment/productivity loss is calculated as the sum of absenteeism and the product of presenteeism and time at work.
Change from baseline in chronic rhinosinusitis symptoms | 6 Months
  Participants will complete the validated 22-item SinoNasal Outcomes Test (SNOT-22) to evaluate change in chronic rhinosinusitis symptoms. Each of the 22 symptoms on the questionnaire are rated by the participant from 0 (no problem) to 5 (bad). A sum of the 22 item scores provides the overall score, which can range from 0 to 110.
Improvement in tympanogram | 6 Months
  Percentage of participants with an abnormal tympanogram (type B or C) at baseline who have a normal (type A) or improved (type B to type C) tympanogram at follow-up.
Improvement in ability to perform a Valsalva maneuver | 6 Months
  Percentage of participants unable to perform the Valsalva maneuver (negative) at baseline who are able to perform the maneuver (positive) at follow-up.
Improvement in tympanic membrane position | 6 Months
  Percentage of participants with a retracted tympanic membrane at baseline who have a normal tympanic membrane position at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Edward D McCoul, MD, PhD, Principal Investigator — Ochsner Health System, New Orleans, LA
Locations (11):
- United States (11):
  - Breathe Clear Institute, Torrance, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Augusta ENT and Allergy, Evans, Georgia
  - St. Vincent Anderson Hospital, Anderson, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ear Nose and Throat Consultants, Southfield, Michigan
  - St Cloud ENT, Saint Cloud, Minnesota
  - ENT Consultants of Nevada, Las Vegas, Nevada
  - Lakeside ENT, Canandaigua, New York
  - National Allergy and ENT, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607